CLINICAL TRIAL: NCT06168279
Title: Assessment of Virtual Digital Articulation Versus Hand-articulation Accuracy for Occlusal Registration in Orthognathic Surgery (Randomized Clinical Trial)
Brief Title: Virtual Digital Articulation Versus Hand-articulation Accuracy for Occlusal Registration in Orthognathic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, abdullah gamal abdullah alawlaqi, phd candidate and principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: omfs 337
Record Dates: First submitted 2023-11-25; First posted 2023-12-13 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2023-12

CONDITIONS: Dentoalveolar Deformities
Keywords: digital occlusal articulation; virtual occlusal registration

STUDY DESIGN:
Intervention Model Description: comparison between conventional occlusal articulation and virtual occlusal articulation for accurate of occlusal registration
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional group (Active Comparator): hand occlusal articulation
  Interventions: Procedure: hand occlusal articulation
- study group (Active Comparator): digital occlusal articulation
  Interventions: Procedure: digital occlusal articulation

INTERVENTIONS:
Procedure: hand occlusal articulation — The upper and lower cast will be scanning separately then will be articulated manually in the final occlusion then scanned after that the stl file will insert to the software to complete virtual planning of orthognathic surgery to made splints that will be using in the operation
  Arms: conventional group
Procedure: digital occlusal articulation — Both upper and lower casts will be scanning separately, then the 3D casts will be articulating by using 3d virtual program to obtained the final occlusion after that the stl file will insert to the software to complete virtual planning of orthognathic surgery to made splints that will be using in the operation
  Arms: study group

SUMMARY:
Conventionally, orthognathic occlusal planning is performed by physically articulating the study models until a well interdigitated occlusion is achieved. this is undertaken in conjunction with the analysis of the face and jaw bones for surgical planning.

Computer-assisted planning now allows digital planning of orthognathic surgery, including assessment of the quality of the final occlusion and printing of the guiding occlusal wafers. This can be achieved through the replacement of the defective images of the dentition produced by the cone beam computed tomography (CBCT) scan with accurate digital images of the study models, captured using CBCT or laser scanning

DETAILED DESCRIPTION:
The determination of an ideal dental occlusion is a vital step in planning orthognathic surgery. Conventionally, a dental occlusion is determined using model surgery based on two dimensional cephalometric planning for the movement of maxillary and mandibular segments. Later, acrylic surgical splints were fabricated in the articulator and used in operating rooms to reposition jaw bones. This conventional method is well established, widely used, and inexpensive. However, its main disadvantages are that patients experience discomfort during the impression procedure, and making dental models and performing model surgery are time consuming. In addition, there is a need for storing dental casts, and errors may occur during this procedure. Computer-aided simulation surgery and three-dimensional planning have become popular. Nadjmi et al. proposed an experimental method for virtual occlusions and demonstrated that the mean distance between their conventional and virtual manual occlusion was small. Adolphs et al. scanned a dental cast and aligned the tooth image for a virtual occlusion by using a software program and reported no difference between the virtual and traditional splint when fitted to a patient's dentition. Wu et al. proposed an experimental haptic simulation framework to determine the virtual occlusion in digital models and showed that the translation and angular deviation of virtual results were smaller compared with the benchmark. However, because the conventional dental impression and model are still required in the computer-aided system and the occlusion setup is determined by the dental model, it cannot be described as fully digital three dimensional planning.

Intraoral digital scanning is an innovative dental technology that has advanced the field of prosthodontics and orthodontics. This technique has been introduced as an alternative to the conventional method for scanning patients' dentition and has become a convenient method for digital impression and model fabrication.The scans can be imported to a software program for planning orthodontic treatment. However, the use of intraoral scanning for the digital setup of the final dental occlusion in three-dimensional orthognathic surgery planning has not yet been reported.

ELIGIBILITY:
Inclusion Criteria:

* Age arrange from 18-40 yr
* Patient requiring orthognathic surgery to correct dentofacial occlusion deformity
* Patient should be free from any significant medical condition that could affect healing or outcomes

Exclusion Criteria:

* • One or more missing central incisors, canines, and/or first molars

  * Patient with facial cleft
  * Patient with significant medical condition

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
accuracy of occlusal registration | immediate after one month of procedure
  The study will be comparing accuracy in occlusal registration ( between peroperative occlusal registration and postoperative occlusal registration ) between the two groups conventional (hand occlusal articulation) and study group (digital virtual occlusal articulation)
  accuracy will be assessed through measuring difference between preoperative and postoperative in software using reference points. measurement will be in millimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Abdullah, Cairo, Egypt